CLINICAL TRIAL: NCT06246981
Title: Evaluation of the Effect of Pelvic Morphology in Quiet Standing on Spatiotemporal Parameters and Pelvic Movements During Gait
Brief Title: Pelvic Morphology in Quiet Posture and Its Effect on Gait
Status: Completed | Type: Observational
Sponsor: Afyonkarahisar Health Sciences University (Other)
Responsible Party: Principal Investigator, Yunus Emre Kundakçı, Asst. Prof., Afyonkarahisar Health Sciences University
Other Study IDs: 2023/9-387
Record Dates: First submitted 2024-01-29; First posted 2024-02-07 (Actual); Last update posted 2025-03-14 (Actual); Status verified 2024-06

CONDITIONS: Anatomy; Morphology; Gait; Pelvis
Keywords: Morphology; Pelvic movement; Pelvis; Posture; Gait

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

SUMMARY:
Pelvic orientations observed in the pelvis during quiet standing position the standard orientation of the pelvis, causing pelvic tilt, pelvic obliquity and pelvic rotation. There is a need to understand the relationship between these orientation disorders and gait. This is because the orientation of the pelvis both in standard standing posture and during gait is an integral part of physiotherapy assessment due to the various problems associated with abnormal pelvic position, including musculoskeletal disorders of the lumbar spine, pelvis, hips and knees. The aim of this study was to describe the morphology of pelvic orientation during static standing posture in an asymptomatic young Turkish population aged 19 to 29 years and to examine the relationship between morphologic changes and changes in pelvic tilt, pelvic obliquity and pelvic rotation angles during gait.

DETAILED DESCRIPTION:
The pelvic bones are the key structures that connect the trunk to the lower extremities, support the body's weight and transfer the load to the lower extremities. The symmetrical orientation of the pelvis about the horizontal plane determines the morphology of the pelvis during static standing posture. When the symmetry of the pelvis is disturbed, its effect on gait parameters is unclear. In clinical practice, the pelvis functionally has 3 basic rotational movements during a gait activity. These are associated with upward (positive) or downward (negative) movement of the pelvis in the coronal plane; forward or backward movement in the sagittal plane; and internal (positive) or external (negative) movement in the horizontal plane. Although these angles are determined by the balance of muscle and ligament forces acting between the pelvis and adjacent segments, they can also be affected by changes in pelvic morphology. If the height of the iliac crest in the coronal plane is significantly different on the right and left, this indicates a pelvic oblique asymmetry. On the other hand, pelvic asymmetries can also be seen in the sagittal plane. Here, the pelvic tilt angles on the right and left are usually significantly different from each other. In the literature, morphologic analyses of the pelvis in static standing posture or dynamically during a gait activity have been performed separately. However, to our knowledge, there is no study on the extent to which pelvic asymmetries seen during gait are affected by the morphology of the pelvis in static standing posture. In this study, the pelvis of young adults aged 19-29 years will be evaluated in two stages. In the first stage, pelvic orientation (pelvic tilt, pelvic obliquity and pelvic rotation) will be measured during static standing using a PALM (palpation meter pelvic inclinometer) inclinometer and leg length will be measured using a tape measure. In the second stage, spatio-temporal parameters and pelvic parallels will be assessed during walking using a wearable inertial sensor. With the data obtained, it is aimed to classify the pelvic morphology of the participants as symmetrical and asymmetrical in the literature and to reveal the effects of pelvis types specific to this classification on the parameters during walking. The results of this study will accurately and precisely measure the orientation of the pelvis with objective tools under static and dynamic conditions, which may increase the reasoning skills and understanding of rehabilitation strategies to be developed for pathologies related to this region. In addition, this study will elucidate the effect of pelvic asymmetries on the kinetic and kinematics of the pelvis on gait quality.

ELIGIBILITY:
Inclusion Criteria:

* 19 to 29 years old
* Not having a confirmed health problem (The participant's use of acute or chronic medication that causes neuromusculoskeletal system disorder will be confirmed by asking)

Exclusion Criteria:

* Syndromes related to the Central Nervous System and/or locomotor system that interfere with proper psychomotor development,
* Disorders potentially causing postural pathologies: genetic syndromes, hormonal disorders, neuromuscular diseases, congenital locomotor system defects,
* Participants with a body mass index over 30,
* Those who did not give written informed consent to participate in the study.

Ages: 19 Years to 29 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Study Population: The participants of the study will consist of young adults between the ages of 19-29 studying at the Faculty of Health Sciences and Atatürk Vocational School of Health Services.
Sampling Method: Non-Probability Sample
Enrollment: 167 (Actual)
Dates: Start 2024-01-20 (Actual); Primary Completion 2024-10-20 (Actual); Study Completion 2025-03-05 (Actual)

PRIMARY OUTCOMES:
Morphological evaluation of the pelvis | Baseline
  A caliper-based inclinometer (PALM palpation meter pelvic inclinometer) will be used to assess pelvic morphology in the standing position. The PALM consists of an inclinometer and two caliper arms. The assessments involve positioning the two calipers of the PALM in contact with the two bony prominences and reading the angle. The iliac crest, anterior superior iliac spine and greater trochanter on each side of the pelvis respectively will be marked by the assessor as reference measurement points. The calipers of the inclinometer will be placed in the horizontal plane on the same reference points left and right. Thus, the following 3 angles between the inclinometer and the horizontal plane will be measured in degrees.
Gait analysis | Baseline
  Gait parameters (gait speed, cadence, double stride length, double stride duration, single support and double support periods, sway and stance phase durations) will be evaluated with the BTS G-Walk device with the 10 Meter Walk Test.

SECONDARY OUTCOMES:
Leg Length Measurement | Baseline
  A standard clinical tape measure that allows 1 mm measurements will be used to measure leg length. Measurements will be taken in the supine position for the right and left extremities. The proximal end of the tape measure will be inserted into the anterior superior iliac spine. Measurements will then be taken by sliding the tape measure from proximal to distal until it collapses under the distal end of the medial or lateral malleolus, respectively

CONTACTS AND LOCATIONS:
Overall Officials: Yunus Emre Kundakcı, Asst. Prof., Principal Investigator — Afyonkarahisar Health Sciences University
Locations (1):
- Afyonkarahisar Health Science University, Afyonkarahisar, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided